CLINICAL TRIAL: NCT06751277
Title: A Single-arm, Open-label, Multi-center Clinical Trial of Iparomlimab and Tuvonralimab (QL1706, Anti-PD-1 /CTLA-4 Combination Antibody) Combined with Chemotherapy in the Treatment of Recurrent or Metastatic Endometrial Cancer
Brief Title: QL1706 Combined with Chemotherapy in the Treatment of Recurrent or Metastatic Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: xiang yang (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, xiang yang, Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-EdC-IIT-001
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Recurrent or Metastatic Endometrial Cancer
Keywords: immunotherapy; anti-PD-1 antibody; anti-CTLA-4 antibody.; endometrial cancer
MeSH Terms: conditions — Recurrence; Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): QL1706（iparomlimab and tuvonralimab a bifunctional MabPair® product of anti-PD-1 IgG4 and anti-CTLA-4 IgG1 antibodies） plus carboplatin and paclitaxel for six to eight cycles at the investigator's discretion, followed by QL1706 until disease progression, development of unacceptable toxicity, lack of benefit as judged by the investigator, withdrawal of consent, completion of 2 years of QL1706 treatment, or other reasons specified in the protocol.
  Interventions: Drug: QL1706 plus carboplatin plus paclitaxel for six to eight cycles at the investigator's discretion, followed by QL1706

INTERVENTIONS:
Drug: QL1706 plus carboplatin plus paclitaxel for six to eight cycles at the investigator's discretion, followed by QL1706 — QL1706 plus carboplatin plus paclitaxel for six to eight cycles at the investigator's discretion, followed by QL1706

SUMMARY:
the investigators planned to evaluate the efficacy and safety of QL1706 in combination with chemotherapy as first-line systemic therapy in approximately 26 patients with newly diagnosed recurrent or metastatic endometrial cancer in a single-arm, open-label, multicenter study.

The main questions it aims to answer are:

Evaluate the efficacy and safety of QL1706 plus chemotherapy as first-line systemic therapy for recurrent or metastatic disease.

According to the treatment regimen, a total of 26 subjects were enrolled. Eligible subjects received QL1706 (5mg/kg, Q3W, d1) plus carboplatin (AUC=5, Q3W, d1) plus paclitaxel (175mg/m2, Q3W, d1) for six to eight cycles at the investigator's discretion, followed by QL1706 (5mg/kg, Q3W, d1). d1) until disease progression, development of unacceptable toxicity, lack of benefit as judged by the investigator, withdrawal of consent, completion of 2 years of QL1706 treatment, or other reasons specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written ICF.
2. The age at enrollment was ≥18 years old, ≤75 years old, female.
3. Eastern Cooperative Oncology (ECOG) performance status of 0 or 1.
4. Expected survival time ≥3 months.
5. Histologically confirmed stage III/IV or recurrent endometrial cancer, who have not received first-line systemic anticancer therapy, and are not suitable for other treatments other than systemic therapy (e.g., unable or unable to tolerate surgery, unsuitable for radiotherapy, etc.).
6. Presence of measurable lesions as required by: a) at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1); Lymph nodes with the long diameter of non-lymph node lesions ≥10mm or the short diameter of lymph node lesions ≥15mm can be measured repeatedly. b) Lesions receiving external beam radiation therapy (EBRT) or locoregional therapy (such as radiofrequency ablation) must show subsequent evidence of substantial size increase to be considered target lesions.
7. Good function of major organs:
8. Female subjects of childbearing potential must undergo a urine or serum pregnancy test within 3 days before the first dose of medication (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test should be performed, and the result is negative). If a female subject of childbearing potential has sex with an unsterilized male partner, the subject must be using an acceptable method of contraception from the time of screening and must agree to continue using contraception for 120 days after the last dose of study drug. Discontinuation of contraception after this time point should be discussed with the investigator.
9. Participants were willing and able to comply with the scheduled visits, treatment protocols, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Participated in treatment with the investigational drug or used the investigational device within 4 weeks before the first dose of QL1706.
2. Enroll in another clinical study at the same time, unless it is the follow-up period of an observational (nonintervention) clinical study or an intervention study (defined as the first dose of the study drug is more than 4 weeks after the last dose of the previous clinical study or more than 5 half-lives of the study drug, whichever is the longest).
3. Carcinosarcoma (malignant mixed Mullerian tumor), endometrial leiomyosarcoma or other high-grade sarcoma, or endometrial stromal sarcoma.
4. Patients with other active malignant tumors within 2 years before enrollment. Exclusions were made for locally curable malignancies that appeared cured, such as squamous cell carcinoma of the basal or skin, superficial bladder cancer, and carcinoma in situ of the cervix or breast.
5. Active autoimmune disease requiring systemic treatment within 2 years before the initiation of study treatment, or autoimmune disease with potential recurrence or planned treatment as judged by the investigator; Exceptions include skin diseases that do not require systemic treatment (e.g., vitiligo, alopecia, psoriasis, or eczema); Hypothyroidism due to autoimmune thyroiditis requires only stable doses of hormone replacement therapy. Well-controlled type I diabetes; Subjects who have had complete remission of childhood asthma without any intervention in adulthood; The investigator judged that the disease would not recur in the absence of an external trigger.
6. Inflammatory bowel disease associated with active disease or requiring clinical management (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
7. History of a known positive test for human immunodeficiency virus or a known positive test for acquired immunodeficiency syndrome.
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
9. Known presence or history of interstitial lung disease.
10. History of gastrointestinal perforation and/or fistula within 6 months before enrollment.
11. The subject had a necrotizing lesion on examination within 4 weeks before enrollment and was judged by the investigator to be at risk for major bleeding.
12. Serious infection within 4 weeks before the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.
13. Known active pulmonary tuberculosis (TB). Subjects suspected to have active TB were examined by chest X-ray, sputum, and excluded by clinical signs and symptoms.
14. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 1000IU/mL, and patients with active hepatitis C should be excluded. Inactive hepatitis B surface antigen (HbsAg) carriers, treated patients with stable hepatitis B (HBV DNA<1000IU/mL), and patients with cured hepatitis C were eligible. For subjects who were positive for HCV Ab, they were eligible to participate in the study only if they had a negative HCV RNA test result.
15. Known presence of leptomeningeal metastases, spinal cord compression, leptomeningeal disease, or active brain metastases. However, subjects with measurable lesions outside the central nervous system were allowed if they: 1) had not been previously treated and were currently asymptomatic (e.g., absence of neurological dysfunction, epilepsy, or other symptoms and signs typical of central nervous system metastases; No need for corticosteroids). 2) treatment-naive asymptomatic patients who have been radiographically stable for at least 4 weeks (e.g., no new or expanding brain metastases) before the initiation of study treatment and who have stopped systemic glucocorticoids and anticonvulsants for at least 2 weeks.
16. Subjects with pleural, pericardial, or ascites that could not be stably controlled by repeated drainage or other methods, as judged by the investigator.
17. Uncontrolled coexisting medical conditions, including symptomatic congestive heart failure (New York Heart Association functional class 3 or 4), uncontrolled hypertension, unstable angina, poorly controlled arrhythmias, evidence of acute or ongoing myocardial ischemia, severe active peptic ulcer disease, or gastritis, Or mental illness/social condition that would limit compliance with study requirements or affect the participant's ability to provide written informed consent. Any arterial thromboembolic event occurred within 6 months before enrollment, including myocardial infarction, cerebrovascular accident, or transient ischemic attack, a history of deep-vein thrombosis, pulmonary embolism, or any other major thromboembolism.
18. Have received immune checkpoint inhibitors (such as anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy, and any treatment targeting tumor immune mechanism.
19. Subjects required systemic treatment with corticosteroids (>10mg prednisone equivalent per day) or other immunosuppressive drugs for 14 days after taking the study drug. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent were allowed. Subjects allowed topical, ocular, intra-articular, intranasal, and inhaled corticosteroids (with minimal systemic absorption). Physiological alternative doses of systemic corticosteroids were allowed, even with >10 mg/day prednisone equivalents. Short-term use of corticosteroids was permitted for prevention (e.g., contrast allergy) or treatment of nonautoimmune conditions (e.g., delayed hypersensitivity from contact allergens).
20. Had undergone major surgical surgery within 30 days (at the discretion of the investigator) before the first dose of QL1706 or had not fully recovered from a previous surgery. Local procedures (e.g., placement of systemic ports, core needle biopsies, and prostate biopsies) were allowed if they were performed at least 24 hours before the first administration of the study treatment.
21. Received the last radiation or antitumor therapy (chemotherapy, targeted therapy, herbal medicine for tumor disease control, or tumor embolization, etc.) within 4 weeks before the first dose of QL1706.
22. Lack of resolution of toxicity from previous antineoplastic therapy was defined as failure to return to NCI CTCAE, version 5.0, grade 0 or 1, or to levels specified in the inclusion/exclusion criteria, with the exception of alopecia. Subjects with irreversible toxicity that is not expected to worsen with study drug administration (e.g., hearing loss) may be enrolled after consultation with the medical monitor. Subjects with long-term radiation-induced toxicity that, in the judgment of the investigator, did not recover from, after consultation with the medical monitor, may be included in the study.
23. Received a live vaccine within 30 days before the first dose of QL1706 or was planned to receive a live vaccine during the study.
24. Known history of severe hypersensitivity reactions to other monoclonal antibodies.
25. Known hypersensitivity to any component of QL1706, carboplatin, or paclitaxel preparations.
26. Pregnant or lactating women.
27. Any condition considered by the investigator to be potentially risky to receive the study drug, or that would interfere with the evaluation of the study drug or the safety of the subjects or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 5 months
  The best overall response (BOR) was defined as the proportion of subjects who achieved a confirmed CR or PR (according to RECIST v1.1).

SECONDARY OUTCOMES:
PFS | up to 13months
  It was defined as the time from the first use of a study drug to documentation of disease progression (according to RECIST v1.1) or death from any cause, whichever occurred first. Subjects who were alive without disease progression at the time of data cutoff for analysis were censored at the last tumor assessment. Subjects who did not undergo postbaseline assessments were censored at the date of the first dose.
DoR | up to 5 months
  It was defined as the time from the first documentation of an objective response (CR or PR) to the first documentation of objective disease progression (according to RECIST v1.1 criteria) or death from any cause, whichever occurred first. Subjects who were alive without disease progression at the time of data cutoff for analysis were censored at the date of the last tumor measurement. DoR was evaluated only in subjects who achieved CR or PR in response.
OS | up to 45 months
  time from first use of a study drug until death from any cause. For those subjects who were alive at the time of data cutoff, censoring will be performed at the last known date of survival. Subjects who did not provide any follow-up information were censored at the date of enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No